CLINICAL TRIAL: NCT05906108
Title: An Integrated WeChat-based Intervention for University Students With Internet Addiction: a Pilot Randomized Controlled Trial
Brief Title: WeChat-based Intervention for Internet Addiction
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Prof. Wang Man-Ping (Other)
Responsible Party: Sponsor-Investigator, Prof. Wang Man-Ping, Professor, The University of Hong Kong
Organization: The University of Hong Kong (Other)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: SF IA
Record Dates: First submitted 2023-06-06; First posted 2023-06-15 (Actual); Last update posted 2025-07-31 (Actual); Status verified 2025-07

CONDITIONS: Internet Addiction
Keywords: Internet addiction; University students; WeChat-based
MeSH Terms: conditions — Internet Addiction Disorder

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group (Experimental): WeChat-based self-initiated learning, personalized and interactive behavioural support
  Interventions: Behavioral: Self-initiated learning; Behavioral: Personalized and interactive behavioural support
- Control group (Active Comparator): General health information
  Interventions: Behavioral: General health information

INTERVENTIONS:
Behavioral: Self-initiated learning — A WeChat Subscription will be created for delivering the intervention. The educational materials involving introduction to internet addiction, the impact of internet addiction and strategies in coping with IA will be posted to the account at the beginning of the intervention. The materials will be prepared in different format including text and video followed by 3 to 5 multiple choice questions (MCQs), and one post for one topic. Relevant materials can be found by typing the keywords in the account or searching under the content list. Participants will be required to follow the account to study the materials at their own pace and complete the MCQs. There will be no limited access to the materials and attempts for MCQs.
  Arms: Intervention group
Behavioral: Personalized and interactive behavioural support — The intervention group will receive 3-month personalized and interactive behavioural support via WeChat, which including regular messages and real-time conversation. The regular messages will cover the generic information about abstinence support, health warnings, benefits of reducing internet time, knowledge reinforcement, goal setting, encouragement and reminders for self-initiated online learning. The messages will be personalised according to baseline demographic characteristics and internet addiction level, and continually adapted to any change in internet behaviours change reported by subjects during the conversations. A total of 19 messages with a tapering schedule. Personalized real-time conversation via WeChat will be available based on participants' demand.
  Arms: Intervention group
Behavioral: General health information — Participants in control group will receive WeChat messages on general health information (similar frequency as the intervention group) and reminders on follow-up surveys via WeChat. Various topics will be involved in the general health information such as healthy diet, sleep management, exercise and mood management.
  Arms: Control group

SUMMARY:
The study aims to design an integrated model which combined self-initiated online learning and personalized interactive behavioral support delivered via WeChat for university students to reduce internet addiction level.

DETAILED DESCRIPTION:
Internet addiction (IA), also described as pathological or problematic internet use, or internet addiction disorders, refers to a pattern of excessive internet use, and it is a new form of behavioral addiction. There are multiple subtypes of IA including excessive online gaming, sexual preoccupations and excessive messages. The excessive use of internet often generates distress or impairments, and evidence showing IA is accompanied by numerous negative impact physically, psychologically and socially such as ADHD, interpersonal sensitivity4, depression and anxiety, family discord, social problems. Pervious study also suggested IA has a significant correlation with academic performance decrement among students, who were considered as a particular vulnerable population being addicted to internet due to easy access to internet, flexible schedule, positive social atmosphere for computer/smartphone use and lack of parental supervision of internet use. IA is a relatively recent and widespread phenomenon. It was estimated 11% Chinese university students were addicted to internet, and an increase in internet use among Chinese children and adolescents was observed amid the COVID-19 epidemic.

IA is believed have some similarities with substance addiction (e.g. smoking, alcohol drinking and drug abuse) as subjects would undergo same symptoms such as depressed, anxious and lonely, affect neurobiology system with common mechanism, and both suffer from substance withdrawal. The interventions for substance addiction have been adopted to treat IA with promising effect including pharmacotherapy, Cognitive Behavior Therapy (CBT), family-based intervention and motivational interviewing, while the treatment for IA has not been standardized yet. In view of the similar characteristics of IA with substance addiction, brief advice and mobile phone-based personalized behavioral support could be feasible to treat IA which has been proven effective in our previous community-based smoking cessation trial, and the COVID-19 epidemic increased the acceptance of mHealth interventions.

The specific objectives are:

1. . To examine the effectiveness of the integrated model in reducing IA in university students;
2. . To assess the acceptability and feasibility of using the model.

ELIGIBILITY:
Inclusion Criteria:

* 1). Currently a full-time university student in HK;
* 2). Aged 18-25 years;
* 3). Internet Addiction Test (IAT) > 50;
* 4). Able to understand and communicate in Chinese;
* 5). Own a smartphone can access internet and proficiency in using WeChat;

Exclusion Criteria:

* 1) Currently participating in other internet addiction controlling projects or services;
* 2) Experiencing psychiatric/psychological diseases or receiving regular psychotropic medication.

Ages: 18 Years to 25 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 120 (Actual)
Dates: Start 2023-03-10 (Actual); Primary Completion 2023-11-30 (Actual); Study Completion 2023-12-30 (Actual)

PRIMARY OUTCOMES:
internet addiction score | at 1-, 3- and 6-month after baseline
  The primary outcome will be the internet addiction score change assessed by Internet Addiction Test (IAT) which is the most valid instrument for IA assessment. The test contains 20 items which rated on a 5 point Likert Scale (1 point refers to rarely, and 5 point refers to always). Score higher than 50 is considered as experiencing occasional or frequent problems because of internet, and the impact on daily life should be aware

SECONDARY OUTCOMES:
Online hours per week | at 1-, 3- and 6-month after baseline
  The daily online hours will be self-estimated and reported. The sum of the online hours will be calculated every 7 days as the total online hours per week.
Sleep time | at 1-, 3- and 6-month after baseline
  The daily sleeping time will be self-estimated and reported.
Physical activity level | at 1-, 3- and 6-month after baseline
  The physical activity will be measured using International Physical Activity Questionnaire.
Self-rated health | at 1-, 3- and 6-month after baseline
  Self-reported health status will be measured using a single-item scale (in general, would you say that your health is excellent, very good, good, fair, or poor?")
Depression and anxiety | at 1-, 3- and 6-month after baseline
  The Patient Health Questionnaire-4 (PHQ-4) will be used to measure depression and anxiety. The 4-item questionnaire consists of a 2-item depression sub-scale and 2-item anxiety sub-scale. The questions are answered on a four-point Likert Scale. The sum of the scores is categorized into normal (0-2), mild (3-5), moderate (6-8) and severe (9-12). The total score of 3 or greater on each sub-scale suggest depression or anxiety, respectively.
Perceived happiness | at 1-, 3- and 6-month after baseline
  A single-item scale (do you feel happy in general?) on an 11-point Likert Scale (0-10) which has been demonstrated valid and reliable in measuring happiness will be used.
Academic performance | at 1-, 3- and 6-month after baseline
  Participant's academic performance will be assessed by " In general, would you say your academic performance is Excellent/Very good/Good/Fair/Poor?

CONTACTS AND LOCATIONS:
Locations (1):
- School of Nursing, The University of Hong Kong, Hong Kong, Please Select, Hong Kong